CLINICAL TRIAL: NCT02138045
Title: A Randomized, Double-blinded, Single-centre, Parallel-group, Placebo-controlled, Prospective Trial of Neuroprotective Effect of Liraglutide for Treatment of Diabetic Neuropathy.
Brief Title: Treatment of Diabetic Neuropathy With Liraglutide
Acronym: TODINELI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Asbjørn Mohr Drewes, Professor, MD, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TODINELI
Record Dates: First submitted 2014-05-13; First posted 2014-05-14 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; Diabetic Neuropathy; Liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo treatment (Placebo Comparator): Placebo solution will be slowly titrated to maximum tolerable dose in order to minimize potential side-effects, hence treatment will follow:
  First and second week: 0.6 mg/day; Third and fourth week: 1.2 mg/day and Fifth and to sixth week: 1.8 mg/day.
  Interventions: Drug: Placebo treatment
- Liraglutide treatment (Active Comparator): Liraglutide will be slowly titrated to maximum tolerable dose in order to minimize potential side-effects, hence treatment will follow:
  First and second week: 0.6 mg/day; Third and fourth week: 1.2 mg/day and Fifth and to sixth week: 1.8 mg/day.
  Interventions: Drug: Liraglutide treatment

INTERVENTIONS:
Drug: Placebo treatment — Treatment continues at highest tolereable dose (minimum 1.2 mg/day). Intervention time 26 weeks at target dose.
  Arms: Placebo treatment
Drug: Liraglutide treatment — Treatment continues at highest tolereable dose (minimum 1.2 mg/day). Intervention time 26 weeks at target dose.
  Arms: Liraglutide treatment

SUMMARY:
The purpose of this trial is to explore whether liraglutide has a long term effect on clinical symptoms and biomarkers in patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Abile person of Northern European descent
* Age between 18 to 65 years
* A verified diagnosis of DM type 1 for minimum 2 years (HbA1C=7%)
* Stable DM treatment (Treatment is considered stable when the patient has been treated with basal-bolus insulin, premixed insulin or continously infused insulin with an insulin dose considered stable by investigator for at least 3 months prior to screening.)
* The participants must be able to read and understand Danish.
* Peripheral diabetic neuropathy ensured by having abnormal nerve conduction velocity
* BMI equal to or above 22
* Personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.
* Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other trial procedures.

Exclusion Criteria:

* Diabetes mellitus type II
* Estimated glomerular filtration rate (s-creatinin/eGRF) < 60 ml/min/1.37m2
* Calcitonin > 25
* HbA1c level < 7%
* Patients with any clinically significant laboratory abnormalities, that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results.
* Patients on GLP-1 receptor agonist treatment (exenatide, liraglutide or others) or pramlintide or any DPP-4 inhibitor within 3 months prior to screening.
* Other neurological and/or psychiatric disease
* Treatment of other endocrinological disease except hypothyreosis
* Malignant neoplasms requiring chemotherapy, surgery, radiation or palliative care in the previous 5 years.
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma.
* Personal history of non-familial medullary thyroid carcinoma
* Known abuse or alcohol and/or medicine (Alcohol use in accordance with the recommendations by the Danish Health and Medicines Authority are allowed).
* Known allergy to liraglutide.
* Participation in other clinical trials less than 3 months prior to inclusion
* Female patients who are pregnant or lactating, or intend to become pregnant and male patients who intend to father a child during course of the study.
* In women, a serum pregnancy test will be conducted at baseline based on h-CG in the blood. The investigator will have to ensure that fertile female patients use a safe contraception method during the study and for at least 15 hours after termination of the study medication period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
RIII withdrawal reflex activity (using standard electromyography) | After 6 months of treatment with Liraglutide
Evoked brain potentials (using standard electroencephalographic brain imaging). | After 6 months of treatment with Liraglutide

SECONDARY OUTCOMES:
Heart rate variability/ alterations in simpatico-vagal balance (24 h Holter monitoring) | After 6 months of treatment with Liraglutide
Resting brain activity (spectral analysis of resting brain activity) | After 6 months of treatment with Liraglutide
Microstructural brain neurodegeneration (assessed by diffuse tensor imaging) | After 6 months of treatment with Liraglutide
Variety in day/night blood pressure | After 6 months of treatment with Liraglutide
Gut transit assessed by SmartPill (pH, pressure and transit in stomach, small and large intestine) | After 6 months of treatment with Liraglutide
Quantitive sensory testing of pressure algometry in muscle | After 6 months of treatment with Liraglutide
Capacity of descending pain inhibition induced by a cold pressor test (2C in 120 sec) | After 6 months of treatment with Liraglutide
Profile of inflammatory cytokines including IL-beta, TNF-alfa, IL6, MCP-1 and specific markers sCD163, sMR, neopterin and HO-1. | After 6 months of treatment with Liraglutide
Metabolic risk factors expressed as adipokines (adiponectin, leptin, resistin) and inflammatory cell markers | After 6 months of treatment with Liraglutide
Self assessed symptomatology (Michigan neuropathy screening tool, Quality of life (SF-36), Pain catastrophizing scale (PCS) and self-assessed gastro-intestinal symptoms (PAGI-SYM)) | After 6 months of treatment with Liraglutide
OCT | After 6 months of treatment with Liraglutide

OTHER OUTCOMES:
HbA1C | After 6 months of treatment with Liraglutide
Biochemical lipid profile | After 6 months of treatment with Liraglutide
Heart rate and blood pressure | After 6 months of treatment with Liraglutide
Weight/body mass index | After 6 months of treatment with Liraglutide

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M. Drewes, Professor, Principal Investigator — Mech-Sense, Department of Medical Gastroenterology, Aalborg Hospital
Locations (1):
- Mech-Sense, Department of Medical Gastroenterology, Aalborg University Hospital, Aalborg, Jutland, Denmark

REFERENCES:
- [Derived] Arendt Nielsen T, Sega R, Uggerhoj Andersen C, Vorum H, Drewes AM, Jakobsen PE, Brock B, Brock C. Liraglutide Treatment Does Not Induce Changes in the Peripapillary Retinal Nerve Fiber Layer Thickness in Patients with Diabetic Retinopathy. J Ocul Pharmacol Ther. 2022 Jan-Feb;38(1):114-121. doi: 10.1089/jop.2021.0055. Epub 2021 Dec 16. PMID 34918951
- [Derived] Nissen TD, Meldgaard T, Nedergaard RW, Juhl AH, Jakobsen PE, Karmisholt J, Drewes AM, Brock B, Brock C. Peripheral, synaptic and central neuronal transmission is affected in type 1 diabetes. J Diabetes Complications. 2020 Sep;34(9):107614. doi: 10.1016/j.jdiacomp.2020.107614. Epub 2020 May 8. PMID 32571684
- [Derived] Nedergaard RB, Nissen TD, Morch CD, Meldgaard T, Juhl AH, Jakobsen PE, Karmisholt J, Brock B, Drewes AM, Brock C. Diabetic Neuropathy Influences Control of Spinal Mechanisms. J Clin Neurophysiol. 2021 Jul 1;38(4):299-305. doi: 10.1097/WNP.0000000000000691. PMID 32501945
- [Derived] Brock C, Hansen CS, Karmisholt J, Moller HJ, Juhl A, Farmer AD, Drewes AM, Riahi S, Lervang HH, Jakobsen PE, Brock B. Liraglutide treatment reduced interleukin-6 in adults with type 1 diabetes but did not improve established autonomic or polyneuropathy. Br J Clin Pharmacol. 2019 Nov;85(11):2512-2523. doi: 10.1111/bcp.14063. Epub 2019 Aug 30. PMID 31338868